CLINICAL TRIAL: NCT02792621
Title: Assessing the Effects of Increased Mitochondrial Function on Skeletal Muscle Performance in Older Men; a Pilot Study
Brief Title: Increasing Mitochondrial Function on Skeletal Muscle Performance in Older Men
Acronym: Rejuvenate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Devon and Exeter NHS Foundation Trust (Other)
Collaborators: University of Exeter (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: R&D no 1608287
Record Dates: First submitted 2016-05-24; First posted 2016-06-07 (Estimated); Last update posted 2020-03-10 (Actual); Status verified 2018-04

CONDITIONS: Impaired Mitochondrial Function, Muscle Performance
MeSH Terms: interventions — acipimox

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- active oral supplement (Experimental): The active supplement will contain the prescription drug Acipimox (250 mgs) , a nicotinic acid precursor traditionally used to lower blood lipid levels. The supplement will be administered 3 times per day, for a 14 day period.
  Interventions: Dietary Supplement: Acipimox
- placebo supplement (Placebo Comparator): The placebo supplement will contain only cellulose microcrystalline. This is an inert substance widely used in many pill and tablet formulations. It is an insoluble fibre and is not absorbed into the blood stream therefore is unlikely to cause toxicity when taken orally.
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: Acipimox — Oral supplement containing Acipimox 250mgs as the active ingredient in blinded label tablet form.
  Arms: active oral supplement
Dietary Supplement: placebo — The placebo supplement will contain only cellulose microcrystalline. This is an inert substance widely used in many pill and tablet formulations. It is an insoluble fibre and is not absorbed into the blood stream therefore is unlikely to cause toxicity when taken orally.
  Arms: placebo supplement

SUMMARY:
As people grow older skeletal muscle gradually becomes smaller and weaker, causing reduced mobility and quality of life. To understand and reverse this negative process investigators need to find new ways of improving the ability of muscle to perform physical activity. There is some evidence that supplements may improve how the mitochondria work, and investigators want to explore this idea in more detail, by measuring how the muscles work and respond to exercise before and after taking the supplement. This will give us the basic information investigators would need to see if this is a useful idea.

DETAILED DESCRIPTION:
A defining feature of ageing is loss of muscle mass ('sarcopenia') and associated functional weakness ('dynapenia'). A common characteristic of dynapenia is lowered mitochondrial content and metabolic function, causing reduced aerobic capacity, increased sensations of effort and impaired lipid oxidation (with resultant glucose intolerance). Exercise training improves mitochondrial and muscle function in ageing populations, however such adaptations remain below that of young counterparts, suggesting alternative approaches are required. Pre-clinical studies show that dietary supplementation with precursors of nicotinamide adenine dinucleotide (NAD+) restore mitochondrial biogenesis and oxidative capacity in ageing rodents and diabetic humans. However, whether NAD+ precursors rejuvenate mitochondrial capacity and, ultimately, muscle function in older humans is unknown. This pilot project will therefore investigate the efficacy of NAD+ precursor supplementation for increasing muscle performance in normally active older men, combined with examination of the molecular and metabolic mechanisms regulating physiological responses.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age between 65-75 years
* Body mass index between 19-29
* No active cardiovascular or metabolic disease
* No active respiratory disease
* No current musculoskeletal injuries
* A sedentary lifestyle (i.e. does not engage in strenuous, planned physical activity)
* The ability to give informed consent

Exclusion Criteria:

* Currently taking a statin drug or NSAIDs
* Have a current peptic ulcer
* Have any renal impairment
* Have a known hypersensitivity to Acipimox

Ages: 65 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-11-08 (Actual); Primary Completion 2018-06-26 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
Change in mitochondrial function | Baseline, day 7, day 14
  Mitochondria will be extracted from muscle samples immediately post-biopsy (biopsies taken baseline, day 7 and day 14) and analysed for content and subsequently for oxidative respiratory function using the Seahorse technique, and maximal rates of Adenosine Triphosphate (ATP) production.

SECONDARY OUTCOMES:
Chronic changes in habitual muscle protein synthetic rates | Baseline and then daily for 14 days
  baseline saliva samples then daily saliva samples following oral ingestion of the stable isotope deuterium oxide (D2O, or 'heavy water') will be analysed by gas-chromatography-pyrolysis-isotope ratio mass-spectrometry analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Etheridge, PhD, Study Director — University of Exeter
Locations (1):
- NIHR Exeter Clinical Research Facility, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No